CLINICAL TRIAL: NCT00586352
Title: Protein Metabolism in Newly Diagnosed Pediatric Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GCRC 1351; IRB 0512-16 (Other: Indiana University)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Protein Metabolism
Keywords: Pediatric; Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal (Active Comparator): Subjects who have normal endoscopic findings
  Interventions: Other: stable isotope infusions
- Newly diagnosed Crohn's disease (Active Comparator): Subjects who are newly diagnosed with Crohn's disease after endoscopy.
  Interventions: Other: stable isotope infusions
- Newly diagnosed Ulcerative Colitis (Active Comparator): Subjects diagnosed with Ulcerative Colitis after endoscopy
  Interventions: Other: stable isotope infusions

INTERVENTIONS:
Other: stable isotope infusions — Subjects receive stable isotope infusions through an IV for about 3 hours. The dosage is based on weight.

SUMMARY:
Inflammatory bowel disease, which includes both Crohn's disease and ulcerative colitis, is a disease of the gastrointestinal tract leading to symptoms of abdominal pain, diarrhea, and growth disturbance. Crohn's disease is a chronic inflammatory process that may affect any part of the gastrointestinal tract, whereas ulcerative colitis is typically present only in the colon. Children with inflammatory bowel disease frequently suffer from disturbances in growth, which may continue into adulthood and result in altered growth outcomes. The metabolic response to inflammatory bowel disease, including increased protein breakdown and decreased protein synthesis may play a significant role in the resulting malnutrition and growth failure from which children with inflammatory bowel disease suffer. The purpose of this study is to compare the rates of protein synthesis within the mucosal lining of the gastrointestinal tract in children Crohn's disease or ulcerative colitis to children who have normal endoscopic examinations. By comparing children with inflammatory bowel disease to normal children, we can begin to determine how alterations in protein metabolism within the lining of the gastrointestinal tract affect whole body protein metabolism, and its consequent effects on growth. In those patients diagnosed with Crohn's disease or ulcerative colitis, a follow-up study will be conducted two weeks following the initiation of steroid therapy to determine its effects on protein metabolism. We hypothesize that children with active inflammatory bowel disease will have increased rates of protein synthesis in the lining of the gastrointestinal tract than patients who have normal endoscopy, and that increases in protein breakdown and protein synthesis will be improved following steroid therapy in children with newly diagnosed inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children between the ages of six and eighteen years of age
* Suspected inflammatory bowel disease or chronic abdominal pain not suspected of having inflammatory bowel disease
* Screening laboratory tests that meet the following criteria (obtained within 4 weeks of enrollment):

  1. Hemoglobin >8.0 g/dL
  2. White blood cell count >3.5 x 109/L
  3. Neutrophils >1.5 x 109/L
  4. Platelets >100 x 109/L
  5. Aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase levels within 3 times the upper limit of normal.
* Parent or guardian signing witnessed, informed consent
* Child (if > age 7) signing assent

EXCLUSION CRITERIA:

* Known malignancy or history of malignancy within 5 years of enrollment.
* Positive stool examination for enteric pathogens including Salmonella and Shigella species, Clostridium difficile, and Giardia lamblia.
* Female subjects who are pregnant, nursing, or planning pregnancy.
* History of substance abuse.
* Poor tolerability of venipuncture or lack of venous access during the study period.
* Inability to comply with study procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Compare gastrointestinal mucosal protein synthesis rates among children with newly diagnosed Crohn's disease and ulcerative colitis to children with normal endoscopic findings. | Week 0

SECONDARY OUTCOMES:
Compare whole body protein metabolism in children with newly diagnosed Crohn's disease and ulcerative colitis before and 2 weeks after initiation of corticosteroid therapy. | Week 0 and Week 2

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Steiner, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University - Riley Hospital for Children, Indianapolis, Indiana, United States